CLINICAL TRIAL: NCT04948554
Title: A Phase 1b Randomized, Double-Blind, Placebo-Controlled, Multiple-Ascending Dose Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of ACE-1334 Plus Standard of Care in Participants With Systemic Sclerosis
Brief Title: A Study of MK-2225 / ACE-1334 in Participants With Systemic Sclerosis With and Without Interstitial Lung Disease (MK-2225-002)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business Reasons
Sponsor: Acceleron Pharma, Inc., a wholly-owned subsidiary of Merck & Co., Inc., Rahway, NJ USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 2225-002; A1334-02 (Other: Acceleronpharma); MK-2225-002 (Other: Merck); 2021-001004-15 (EudraCT Number)
Record Dates: First submitted 2021-06-04; First posted 2021-07-02 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Systemic Sclerosis With and Without Interstitial Lung Disease
Keywords: Diffuse Systemic Sclerosis; Scleroderma; Systemic Sclerosis; Systemic Sclerosis-associated Interstitial Lung Disease
MeSH Terms: conditions — Scleroderma, Diffuse; Scleroderma, Systemic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- Cohort 1: MK-2225 (Experimental): Participants in Cohort 1 will receive MK-2225 at 0.25 mg/kg once every two weeks (Q2W) plus standard of care (SOC) for 12 weeks.
  Interventions: Biological: MK-2225
- Cohort 1: Placebo (Placebo Comparator): Participants in Cohort 1 will receive placebo Q2W plus SOC for 12 weeks.
  Interventions: Biological: Placebo
- Cohort 2: MK-2225 (Experimental): Participants in Cohort 2 will receive MK-2225 at 0.5 mg/kg (or lower) Q2W plus SOC for 12 weeks.
  Interventions: Biological: MK-2225
- Cohort 2: Placebo (Placebo Comparator): Participants in Cohort 2 will receive placebo Q2W plus SOC for 12 weeks.
  Interventions: Biological: Placebo
- Cohort 3: MK-2225 (Experimental): Participants in Cohort 3 will receive MK-2225 at 1.0 mg/kg (or lower) Q2W plus SOC for 12 weeks.
  Interventions: Biological: MK-2225
- Cohort 3: Placebo (Placebo Comparator): Participants in Cohort 3 will receive placebo Q2W plus SOC for 12 weeks.
  Interventions: Biological: Placebo
- Cohort 4: MK-2225 (Experimental): Participants in Cohort 4 will receive MK-2225 at ≤2.0 mg/kg Q2W if needed plus SOC for 12 weeks.
  Interventions: Biological: MK-2225
- Cohort 4: Placebo (Placebo Comparator): Participants in Cohort 4 will receive placebo Q2W plus SOC for 12 weeks.
  Interventions: Biological: Placebo
- Cohort 5: MK-2225 (Experimental): Participants in Cohort 5 will receive MK-2225 (no more frequent than Q2W) ≤2.25 mg/kg Q2W or ≤4.5 mg/kg Q4W if needed plus SOC for 12 weeks.
  Interventions: Biological: MK-2225
- Cohort 5: Placebo (Placebo Comparator): Participants in Cohort 5 will receive (no more frequent than Q2W) placebo plus SOC for 12 weeks.
  Interventions: Biological: Placebo
- Cohort 6: MK-2225 (Experimental): Participants in Cohort 6 will receive MK-2225 (no more frequent than Q2W) ≤2.25 mg/kg Q2W or ≤4.5 mg/kg Q4W if needed plus SOC for 12 weeks.
  Interventions: Biological: MK-2225
- Cohort 6: Placebo (Placebo Comparator): Participants in Cohort 6 will receive (no more frequent than Q2W) placebo plus SOC for 12 weeks.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: MK-2225 — Administered Subcutaneously (SC)
  Other Names: ACE-1334
  Arms: Cohort 1: MK-2225; Cohort 2: MK-2225; Cohort 3: MK-2225; Cohort 4: MK-2225; Cohort 5: MK-2225; Cohort 6: MK-2225
Biological: Placebo — Administered SC
  Arms: Cohort 1: Placebo; Cohort 2: Placebo; Cohort 3: Placebo; Cohort 4: Placebo; Cohort 5: Placebo; Cohort 6: Placebo

SUMMARY:
The purpose of the MK-2225-002 (A1334-02) study is to evaluate the safety and tolerability of MK-2225 (ACE-1334) plus standard of care (SOC) in participants with Systemic Sclerosis (SSc) following multiple doses.

ELIGIBILITY:
The main inclusion and exclusion criteria include but are not limited to the following:

Inclusion Criteria:

* Participants must have SSc, as defined using the 2013 American College of Rheumatology/European League Against Rheumatism criteria
* If participant is on a non-excluded immunosuppressive therapy (e.g. mycophenolate, methotrexate, azathioprine, etc.) the dose should be stable for > 2 months at the time of screening
* Women of childbearing potential must:

  * If sexually active, have used, and agree to use, highly effective contraception without interruption, for at least 28 days prior to starting investigational product, during the study (including dose interruptions), and for 17 weeks (119 days) after discontinuation of study treatment
  * Refrain from breastfeeding a child or donating blood, eggs, or ovum for the duration of the study and for at least 17 weeks (119 days) after the last dose of study treatment
* Male participants must:

  * Agree to use a condom, defined as a male latex condom or nonlatex condom NOT made out of natural (animal) membrane (e.g., polyurethane), during sexual contact with a pregnant female or a female of childbearing potential while participating in the study, during dose interruptions, and for at least 17 weeks (119 days) following investigational product discontinuation, even if he has undergone a successful vasectomy
  * Refrain from donating blood or sperm for the duration of the study and for 17 weeks (119 days) after the last dose of study treatment
* Must agree to not participate in any other study of investigational drugs/devices while enrolled in this study

Exclusion Criteria:

* Participant with SSc-pulmonary arterial hypertension (PAH) (except those participants with mild PAH on up to 2 oral drugs and mean pulmonary arterial pressure < 30 mmHg or low risk by risk calculator)
* In the opinion of the investigator, other clinically significant pulmonary abnormalities (such as obstructive lung disease, asthma, etc.)
* Other investigational therapy received within 1 month or 6 half-lives (whichever is greater) prior to the Screening Visit
* Prior exposure to MK-2225 or other TGF-β antibodies or any TGF-β family targeted biologic or hypersensitivity to the components of MK-2225
* Hypersensitivity to placebo or any of its components
* Previous hematopoietic stem cell transplantation (HSCT) or HSCT planned within the next year
* Major surgical procedures planned during the study period
* Oral prednisone or equivalent > 10 mg/day
* Participant with history of gastric antral vascular ectasia or gastrointestinal bleed
* On anticoagulation therapy (such as prophylaxis anticoagulation, warfarin, direct thrombin inhibitors or other including low molecular weight subcutaneous or intravenous therapeutic heparin), or antiplatelet therapy including aspirin. Use of fish oil supplements within 2 weeks prior to randomization and throughout study is not permitted.
* History of any other medical condition that might interfere with a participant's ability to participate in the study
* Active clinically significant viral, bacterial, or fungal infection, or any episode of infection requiring hospitalization within 4 weeks prior to screening
* Use of cyclophosphamide ≤ 6 months from screening
* Use of nintedanib or pirfenidone ≤ 28 days from screening
* Recent scleroderma renal crisis < 6 months before screening
* Use of tocilizumab ≤ 2 months from screening
* Has received any nonlive vaccine starting from 14 days prior to study intervention or is scheduled to receive any nonlive vaccine through 30 days following study intervention. Exception: COVID-19 vaccine may be administered.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2023-03-10 (Actual); Primary Completion 2023-10-18 (Actual); Study Completion 2023-10-18 (Actual)

PRIMARY OUTCOMES:
Number of Participants with ≥1 Adverse Event (AE) | Up to 20 Weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants who experienced an AE will be reported.
Number of Participants Discontinuing from Study Therapy Due to AE | Up to 12 Weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants who discontinued study treatment due to an AE will be reported.

SECONDARY OUTCOMES:
Area Under the Concentration-Time Curve (AUC0-tau) of MK-2225 | Up to 12 Weeks
  AUC0-tau is the area under the concentration-time curve. Blood samples will be collected at designated timepoints to determine AUC0-tau of MK-2225.
Serum Maximum Concentration (Cmax) of MK-2225 | Up to 12 Weeks
  Cmax is the maximum concentration of the drug observed in plasma. Blood samples will be collected at designated timepoints to determine Cmax of MK-2225.
Time to peak Serum Concentration (Tmax) of MK-2225 | Up to 12 Weeks
  Tmax is the amount of time required to reach Cmax. Blood samples will be collected at designated timepoints to determine Tmax of MK-2225.
Serum Apparent Terminal Half-Life (t1/2) of MK-2225 | Up to 12 Weeks
  t1/2 is the time required for 50% of drug to be cleared from serum. Blood samples will be collected at designated timepoints to determine t1/2 of MK-2225.
Accumulation ratio of AUCtau (RAUC) | Up to 12 Weeks
  RAUC is the accumulation ratio of AUCtau after multiple doses relative to after a single dose. Blood samples will be collected at designated timepoints to determine RAUC of MK-2225.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (16):
- United States (11):
  - UCSD Altman Clinical and Translational Research Institute (Site 1013), La Jolla, California
  - Keck Medical Center ( Site 1001), Los Angeles, California
  - Georgetown University Medical Center ( Site 1010), Washington D.C., District of Columbia
  - University of Florida ( Site 1002), Gainesville, Florida
  - Central Florida Pulmonary Group ( Site 1005), Orlando, Florida
  - Medster Research, LLC ( Site 1017), Valdosta, Georgia
  - University of Kansas Medical Center ( Site 1007), Kansas City, Kansas
  - The Cleveland Clinic Foundation ( Site 1003), Cleveland, Ohio
  - Penn State Milton S Hershey Medical Center ( Site 1004), Hershey, Pennsylvania
  - West Tennessee Research Institute ( Site 1012), Jackson, Tennessee
  - Metroplex Clinical Research Center ( Site 1018), Dallas, Texas
- Mount Sinai Hospital ( Site 1101), Toronto, Ontario, Canada
- Italy (2):
  - Azienda Ospedaliero Universitaria Careggi (Site 1401), Florence, Tuscany
  - Azienda Ospedaliera Universitaria Integrata Di Verona ( Site 1402), Verona, Veneto
- Switzerland (2):
  - Kantonsspital St. Gallen (Site 1301), Sankt Gallen, Canton of St. Gallen
  - Hôpital Neuchatelois ( Site 1304), Neuchâtel, Neuchâtel (fr)

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/